CLINICAL TRIAL: NCT04810013
Title: Noninvasive Measurement of the Cerebral Autoregulation in Neonates and Infants With Complex Congenital Heart Disease After Cardiac Surgery With Cardiopulmonary Bypass at the Pediatric Intensive Care Unit (PICU)
Brief Title: Noninvasive Measurement of the Cerebral Autoregulation in Neonates and Infants With Complex Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: CAR_FN_01
Record Dates: First submitted 2021-02-25; First posted 2021-03-22 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2022-05

CONDITIONS: Complex Congenital Heart Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: non-invasive measurement of cerebral autoregulation — Non-invasive measurement of the cerebral autoregulation in the postoperative period in 80 neonates and infants with complex congenital heart disease undergoing cardiopulmonary bypass surgery. A continuous, moving Pearson's correlation coefficient will be calculated between the arterial pressure and near-infrared spectroscopy signals and displayed continuously during surgery using a laptop computer and the ICM+ software (Cambridge Enterprise).

SUMMARY:
Feasibility of non-invasive cerebral autoregulation measurement at the PICU and impact of changes in oxygen supply

DETAILED DESCRIPTION:
Cerebral protection is a major issue in the treatment of neonates and infants with complex congenital heart disease, because most common long-term morbidities of newborn heart surgery are related not to the heart, but instead to the cognitive challenges experienced by this population. Disruption of cerebral autoregulation in the postoperative period may contribute to brain injury in these patients. Blood pressure management, respirator management and red blood cell transfusion management after cardiopulmonary bypass surgery using endpoints such cerebral autoregulation monitoring might provide a method to optimize organ perfusion and improve neurologic outcome from cardiac surgery in the vulnerable postoperative period.

Primary Objectives: Feasibility of non-invasive cerebral autoregulation measurement at the PICU: Identification of the range of mean arterial blood pressure (MAP) with optimal vasoreactivity (MAPOPT), indicating intact cerebral autoregulation.

Secondary Objectives: Impact of decreased oxygen delivery, increased cerebral oxygen extraction, decreased cardiac output, arterial hypotension, severe hypoxemia and/or severe anemia on cerebral autoregulation.

ELIGIBILITY:
Inclusion Criteria:

* term (37-42 weeks gestation) newborns
* pre- or postnatally diagnosed critical congenital heard disease (CHD)
* admitted to the pediatric cardiac intensive care unit at the Children's Hospital of Tübingen

Exclusion Criteria:

* birth weight <2 kg
* history of neonatal depression (5-min APGAR<5, cord blood pH<7.0, sepsis, or birth asphyxia)
* perinatal seizures
* evidence of end-organ injury
* preoperative cardiac arrest
* significant preoperative intracerebral hemorrhage such as grade 3 or 4 intraventricular hemorrhage.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Range of mean arterial blood pressure | 4within 8 hours after cardiac surgery at the PICU
  Measurement of the range of mean arterial blood pressure (MAP) with optimal vasoreactivity (MAPOPT)

SECONDARY OUTCOMES:
Detection of severe brain injury | before surgery, 12 hours, 48 hours, 72 hours post surgery and before discharge
  Detection of cerebral haemorrhage grade III or IV, cystic periventricular leukomalacia, cerebellar haemorrhage, post-haemorrhagic ventricular dilatation or cerebral atrophy) on routinely performed serial cranial ultrasound scans
Neurological outcome measure | at age of 2 years
  Landmarks of development score (Grenzsteine der Entwicklung Score) aus (Monatsschr Kinderheilkd_2013 · 161:898-910_· DOI 10.1007/s00112-012-2751-0 © Springer-Verlag Berlin Heidelberg 2013 R._Michaelis_· R._Berger_· U._Nennstiel-Ratzel_· I._Krägeloh-Mann Validierte und teilvalidierte Grenzsteine der Entwicklung).
  The score uses dichotomous questions, that asks for a Yes/No response. The score consists of a total of 16 questions, the more questions answered yes, the better the outcome and vice versa. Minimum value is n=0 yes and n=16 no answers, maximum value is n=16 yes and n=0 no answers.
Influence of changed fractional cerebral oxygen extraction (cFTOE) on cerebral autoregulation | within 8 hours after cardiac surgery at the PICU
  Analysis of the influence of changed fractional cerebral oxygen extraction (cFTOE) on cerebral autoregulation.Association between cFTOE and cerebral autoregulation indices (COx and HVx).
Influence of changed arterial blood pressure on cerebral autoregulation | within 8 hours after cardiac surgery at the PICU
  Analysis of the influence of changed arterial blood pressure on cerebral autoregulation. Association between arterial blood pressure (mmHg) and cerebral autoregulation indices (COx and HVx).
Influence of changed arterial oxygen saturation on cerebral autoregulation | within 8 hours after cardiac surgery at the PICU
  Analysis of the influence of changed arterial oxygen saturation on cerebral autoregulation. Association between arterial SPO2 (%) and cerebral autoregulation indices (COx and HVx).
Influence of changed blood hemoglobin concentration on cerebral autoregulation | within 8 hours after cardiac surgery at the PICU
  4. Analysis of the influence of changed blood hemoglobin concentration on cerebral autoregulation. Association between arterial hemoglobin value (g/dL) and cerebral autoregulation indices (COx and HVx).

CONTACTS AND LOCATIONS:
Overall Officials: Felix Neunhoeffer, Principal Investigator — University Children's Hospital Tübingen
Locations (1):
- Univeristy Children's Hospital, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No